CLINICAL TRIAL: NCT03696368
Title: Understanding Diverse Contributors to Gestational Diabetes Mellitus and Its Near-to-Long Term Consequences: An Indiana University Grand Challenges Precision Health Initiative Cohort Study (The Hoosier Moms Cohort)
Brief Title: The Hoosier Moms Cohort
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Haas, Professor of Obstetrics & Gynecology, Indiana University
Other Study IDs: 1808964513
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related; Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal blood
  * Maternal urine
  * Maternal stool
  * Cord blood
  * Infant buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Hoosier Moms Cohort (HMC) study's goal is to better understand the pathophysiology underlying the development of gestational diabetes mellitus (GDM) in pregnant women and its transition to Type 2 diabetes mellitus in mothers and their exposed children.

The HMC study wants to determine what biomarkers (genetic, blood based and behavioral/interventional) can be identified in pregnant women affected with GDM and how those biomarkers can be used to impact preventative care.

DETAILED DESCRIPTION:
Predictive GDM genetic risk models will be tested and refined in the Hoosier Moms Cohort. In addition to prospectively using genetic information to predict GDM risk, the Hoosier Moms Cohort will incorporate the use of wearable/digital devices for collection of detailed behavioral information, support development of novel dietary capture methods, and enable the collection of specimens specifically aimed at multiple 'omics' techniques to engage in a detailed, multidimensional assessment of pathophysiologic pathways and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Gestational age ≤ 20+0 confirmed via American Congress of Obstetrics and Gynecology (ACOG) ultrasound dating guidelines
* 18 years old or greater at time of consent

Exclusion Criteria:

* Pre pregnancy diagnosis of Type 1 Diabetes or Type 2 Diabetes or Screening Hemoglobin A1C that is greater than or equal to 6.5% or two abnormal values on a 3 hours Oral Glucose Tolerance Test (100g load) before 20 weeks gestation
* Pre pregnancy chronic usage of systemic steroids (inhaled and short term usage acceptable)
* Planned pregnancy termination
* Unable to provide informed consent in English or Spanish
* Major fetal anomalies as listed below that are known prior to enrollment. If these are discovered after enrollment, the participant may be allowed to participate, unless the discovered fetal anomaly is a lethal anomaly.

Major Fetal Anomalies to be Excluded:

* Congenital diaphragmatic hernia
* Congenital cystic adenomatoid malformation
* Pleural effusions
* Chylothorax
* Bronchogenic cyst
* Bronchopulmonary sequestration
* Anomalous pulmonary venous return
* Tricuspid atresia
* Mitral atresia
* Double right ventricle
* Ebstein's malformation
* Pulmonary atresia
* Hypoplastic left heart syndrome
* Aortic coarctation
* Fetal arrhythmias (tachycardia or bradycardia)
* Transposition of the great vessels
* Tetrology of Fallot
* Double outlet right ventricle
* Aortic stenosis
* Holoprosencephaly
* Anencephaly
* Dandy-Walker malformation or variant
* Septo-optic dysplasia
* Neural tube defect
* Vein of Galen aneurysm
* Bilateral renal agenesis
* Cystic renal disease (polycystic or multicystic)
* Any genitourinary lesion accompanied by oligohydramnios at <24 weeks
* Obstructive uropathy
* Horseshoe kidney
* Megacystis microcolon
* Achondrogenesis
* Thanatophoric dysplasia
* Thoracic dysplasia
* Osteogenesis imperfect
* Short rib polydactyly
* Any skeletal defect associated with small thorax
* Hypophosphatemia
* Any karyotypic abnormality
* Any suspected genetic syndrome
* Cleft lip/palate
* Micrognathia
* Hydrops
* Fetal anemia (<35% on cordocentesis)
* Neck mass
* Gastroschisis
* Omphalocele

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 pregnant women with an enhanced risk of GDM will be recruited from obstetrical clinics associated with the Indiana University School of Medicine or by self referral.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
GDM Diagnosis | 42 weeks or less gestational age
  Number of subjects diagnosed with GDM

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, MS, Principal Investigator — Indiana University
Locations (6):
- United States (6):
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - IUH Coleman Center for Women, Indianapolis, Indiana
  - IUH Prenatal Diagnosis Clinic, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Tri-state Perinatology at The Women's Hospital, Newburgh, Indiana
  - Women's Health Care PC, Newburgh, Indiana